CLINICAL TRIAL: NCT06195709
Title: ECLECTIC: EstroTEP and Circulating Biomarkers to Determine the Optimal Second Line Therapy for ER-positive HER2-negative Metastatic Breast Cancer Patients
Brief Title: ECLECTIC: EstroTEP and Circulating Biomarkers for ER-positive HER2-negative Metastatic Breast Cancer Patients
Acronym: ECLECTIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Zionexa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2022-12; 2023-506282-66-00 (Registry Identifier: EU trial number)
Record Dates: First submitted 2023-12-07; First posted 2024-01-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
Keywords: Metastatic; PET/CT 18F-FES; Circulating markers
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized, multicentric, open-label, phase III trial conducted in patients with ER+ HER2- metastatic breast cancer progressing on first line treatment with CDK4/6 inhibitor and aromatase inhibitor, and which aims at evaluating the combined value of 18F-FES PET/CT and circulating biomarkers to guide second line treatment decision between investigator's choice second line endocrine therapy (with or without targeted therapy) and chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Endocrine therapy (Sham Comparator): 1. Patients in whom all tumor sites display a FES SUVmax ≥2 AND who have low levels of circulating tumor biomarkers will be treated with endocrine therapy.
  2. Patients in whom 18F-FES PET shows an heterogenous uptake, with one or maximum two tumor sites with low FES uptake (SUVmax <2) that represent less than 20% of all tumor sites and are deemed accessible to local treatment (e.g. stereotactic radiation therapy or another equivalent local therapy) will be treated, if they have low levels of circulating tumor biomarkers, by 2nd line endocrine therapy in Arm A, combined with the local treatment of FES-negative lesions.
  Interventions: Combination Product: Endocrine therapy; Combination Product: Endocrine therapy combined with the local treatment of FES-negative lesions
- Arm B: Chemotherapy (Active Comparator): All other patients, i.e. (i) patients in whom most or ≥3 lesions display a FES SUVmax <2 that are not amenable to local treatment, (ii) patients with high levels of circulating tumor biomarkers, will be randomized between chemotherapy in Arm B and endocrine therapy in Arm C.
  Interventions: Combination Product: Endocrine therapy; Combination Product: Chemotherapy
- Arm C: Endocrine therapy (Active Comparator): All other patients, i.e. (i) patients in whom most or ≥3 lesions display a FES SUVmax <2 that are not amenable to local treatment, (ii) patients with high levels of circulating tumor biomarkers, will be randomized between chemotherapy in Arm B and endocrine therapy in Arm C.
  Interventions: Combination Product: Endocrine therapy; Combination Product: Chemotherapy

INTERVENTIONS:
Combination Product: Endocrine therapy — Consist in single agent endocrine therapy or in combination with targeted therapy, per guidelines and label. LH-RH agonist will be used in combination with endocrine therapy whenever appropriate and per label.
  Other Names: Standardized endocrine therapy regimen
Combination Product: Endocrine therapy combined with the local treatment of FES-negative lesions — Consist in single agent endocrine therapy or in combination with targeted therapy, per guidelines and label. LH-RH agonist will be used in combination with endocrine therapy whenever appropriate and per label. Cases with only 1 or 2 FES-negative lesions that are accessible to local treatment will be reviewed by the Centralized Reading Committee (including a radiation oncologist) to confirm the feasibility of local treatment.
  Other Names: Standardized endocrine therapy regimen
  Arms: Arm A: Endocrine therapy
Combination Product: Chemotherapy — Consist in single agent chemotherapy, poly-chemotherapy, or antibody-drug conjugates, per guidelines and label. Patients who are eligible (per drug label) may receive PARP inhibitor if allocated to Arm B.
  Other Names: Standardized chemotherapy regimen
  Arms: Arm B: Chemotherapy; Arm C: Endocrine therapy

SUMMARY:
Eclectic is a strategy trial; once the class of treatment (endocrine therapy or chemotherapy) has been allocated according to 16α-18F-fluoro-17β-oestradiol (18F-FES) Positron Emission Tomography/Computed Tomography (PET/CT) results and circulating tumor biomarkers, clinicians will decide which treatment to use.

DETAILED DESCRIPTION:
All patients deemed eligible for a second line endocrine therapy will undergo a 18F-FES PET/CT scan and circulating tumor biomarkers assessment (circulating tumor cells (CTC) and, if not available, circulating tumor DNA (ctDNA)). All 18F-FES PET/CT scan will be anonymized and reviewed centrally, and compared to the 18Fluorodeoxyglucose (18F-FDG) PET/CT results before treatment initiation; circulating biomarkers status will be assessed centrally and will remain blinded to investigator and patients.

Endocrine therapy in Arm A and C may consist in single agent endocrine therapy or in combination with targeted therapy. Luteinizing Hormone-Releasing Hormone (LH-RH) agonist will be used in combination with endocrine therapy whenever appropriate and per label. Chemotherapy in Arm B may consist in single agent chemotherapy, poly-chemotherapy, or antibody-drug conjugates. Patients who are eligible (per drug label) may receive Poly-adenosine-5'-diphosphate-ribose Polymerase (PARP) inhibitor if allocated to Arm B.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic invasive breast carcinoma of no special type.
2. Females and males of age ≥18 years.
3. Life expectancy > 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
5. Estrogen Receptor (ER)-positive (≥10%) and HER2-negative (ASCO/College of American Pathologists guidelines) breast cancer, per local assessment on the most recent breast cancer tissue examined.
6. Tumor block Formalin-Fixed Paraffin-Embedded (primary tumor or metastasis) available.
7. Patients whose disease has progressed on first line endocrine therapy with aromatase inhibitor and CDK4/6 inhibitor and who are deemed eligible, per investigator assessment, to a second line endocrine therapy. The progression on first line endocrine therapy with aromatase inhibitor and CDK4/6 inhibitor must have occurred after more than 6 months on treatment.
8. Patients with available 18F-FDG PET/CT imaging
9. Evaluable disease per RECIST criteria and measurable disease per PERCIST criteria.
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and any protocol-related procedures including screening evaluations.
11. Signed informed consent.
12. Patient affiliated to a social security system.

Exclusion criteria:

1. Other breast cancer subtype (e.g. invasive lobular breast carcinoma).
2. One or more prior line of chemotherapy in the metastatic setting.
3. Any other systemic treatment given at metastatic disease than the first line therapy with aromatase inhibitor and CDK4/6 inhibitor.
4. Visceral crisis, per investigator's assessment.
5. Liver-only metastases.
6. Prior exposure to any authorized or experimental agent degrading the estrogen receptor (fulvestrant, oral SERDs, PROTAC, etc).
7. Pregnancy or lactation period.
8. In women of childbearing potential or premenopausal women or women with amenorrhea of less than 12 months, without adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization; LH-RH agonist cannot be considered as an efficient contraceptive measure), positive urinary or serum pregnancy test 72 hours before 18F-FES PET/CT.
9. Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease. Patients with a history of CNS metastases or cord compression are eligible if they have been treated with local therapy (e.g., radiotherapy, stereotactic surgery) and are clinically stable and off anticonvulsants and steroids for at least 4 weeks before treatment start.
10. History of previous cancer or hematological malignancy within 3 years preceding patient enrollment in the trial. Multiple primary breast cancers (controlateral/ipsilateral cancers/local relapses) are allowed pending all tumors were ER+ HER2-.
11. Persons deprived of their freedom or under guardianship or incapable of giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2028-09-27 (Estimated); Study Completion 2029-09-27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 54 months
  PFS is defined as the time from randomization to progression (per RECIST 1.1) or death, among randomized patients.

SECONDARY OUTCOMES:
Progression-Free survival (PFS) | 54 months
  PFS is defined as the time from randomization to progression (per PERCIST 1.0) or death, among randomized patients with available Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) evaluation.
Overall survival (OS) | 54 months
  OS is defined as the time from the date of randomization to the date of death due to any cause, among randomized patients (arms B and C)
Objective response rate (ORR) | 54 months
  ORR is defined as the proportion of patients who have achieved complete response (CR) or partial response (PR) based on local investigator assessment, among randomized patients with measurable disease at baseline,
Clinical benefit rate (CBR) | 24 weeks
  CBR at 24 weeks is defined as the proportion of randomized patients who have achieved either a confirmed complete or partial response, or stable disease for at least 24 weeks after treatment start based on local investigator assessment.
Efficacy criteria: PFS at 24 weeks | 24 weeks
  PFS at 24 weeks will be evaluated in patients allocated to arm A.
Efficacy criteria: OS at 24 weeks | 24 weeks
  OS at 24 weeks will be evaluated in patients allocated to arm A.
Efficacy criteria: ORR at 24 weeks | 24 weeks
  ORR at 24 weeks will be evaluated in patients allocated to arm A.
Efficacy criteria: CBR at 24 weeks | 24 weeks
  CBR at 24 weeks will be evaluated in patients allocated to arm A.
Safety and toxicity and their relationship to study treatment | 54 months
  Incidence, nature and severity of adverse events (AEs) graded according to NCI CTCAE v5.0
EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) after 2 months of treatment | 2 months
  Questionnaire to measure physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items range from 0 to 100. A higher score represents better function and a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Le GOUILL, PhD, Study Director — Institut Curie
Locations (13):
- France (13):
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut du Cancer Montpellier, Montpellier
  - Centre Antoine lacassagne, Nice
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - Bruno MAUCHERAT, Saint-Herblain
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).